CLINICAL TRIAL: NCT04684511
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Phase III Study With a Long-Term, Open-Label Extension to Evaluate the Efficacy and Safety of TRM-201 (Rofecoxib) in Patients With Hemophilic Arthropathy
Brief Title: Rofecoxib Efficacy and Safety Evaluation Trial in Hemophilic Arthropathy
Acronym: RESET-HA
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Low enrollment. The termination of the trial was not based on any safety concerns in the study.
Sponsor: Tremeau Pharmceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TRM-201-HA-301
Record Dates: First submitted 2020-12-21; First posted 2020-12-24 (Actual); Last update posted 2022-10-27 (Actual); Status verified 2022-08

CONDITIONS: Hemophilic Arthropathy
Keywords: Hemophilia; Pain; HA; Joint Pain
MeSH Terms: conditions — Hemophilia A; Pain; Arthralgia | interventions — rofecoxib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TRM-201 (Rofecoxib) (Experimental): 1 TRM-201 tablet taken orally once daily for 12 weeks in Part I and orally once daily for an additional 52 weeks in Part II
  Interventions: Drug: TRM-201 (Rofecoxib)
- Placebo (Placebo Comparator): 1 placebo tablet (to match TRM-201) taken orally once daily for 12 weeks in Part I and then 1 TRM-201 tablet taken orally once daily for an additional 52 weeks in Part II
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TRM-201 (Rofecoxib) — Eligible patients will be randomized to receive TRM-201 or placebo
  Other Names: Placebo
  Arms: TRM-201 (Rofecoxib)
Drug: Placebo — Matching Placebo
  Arms: Placebo

SUMMARY:
This is a multicenter, randomized, double-blind study to evaluate the efficacy and safety of TRM-201 (rofecoxib) versus Placebo in the treatment of patients with hemophilic arthropathy (HA) over a 12-week period (Part I) that is followed by a year-long (52 week) open-label extension (Part II) to further evaluate the safety and maintenance of efficacy of TRM-201.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hemophilia A or B
* Either on a stable prophylaxis regimen for their bleeding disorder (factor, bypassing agent, or nonfactor product therapy) OR currently taking or agree to initiate a gastroprotective agent (esomeprazole) for the duration of the trial
* Diagnosis of Hemophilic Arthopathy for at least 6 months prior to screening
* Chronic symptomatic pain in one or more joint(s) on 20 of the 30 days prior to screening.
* Able and willing to wash out of non-study analgesic medications/agents for at least 7 days prior to Randomization including: acetaminophen (paracetamol), NSAIDs, opioids, cannabinoids, topical analgesics, benzodiazepines, gabapentin/pregabalin-containing products and other antiepileptic drugs used for pain
* Primary source of pain is due to Hemophilic Arthropathy

Exclusion Criteria:

* Taking opioids for greater than 4 days per week prior to screening
* Has a history of advanced renal disease or severe liver disease (within the last 6 months)
* Receiving emicizumab while also receiving activated prothrombin complex concentrate (FEIBA)
* Uncontrolled or poorly controlled hypertension
* History of major cardiac or cerebrovascular disease
* History of an upper GI perforation, obstruction, or major GI bleed or current evidence of GI bleeding
* Has active hepatitis C or hepatitis B infection or uncontrolled HIV. Note: Patients who are HIV positive are allowed to participate if considered to be controlled.
* Has a positive drug screen for all prohibited drugs of potential abuse at screening
* Has had an intra-articular injection (within 3 months), initiated physical therapy (within 30 days) or has had orthopedic surgery (within 4 months) prior to screening

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2022-09-28 (Actual); Study Completion 2022-09-28 (Actual)

PRIMARY OUTCOMES:
The change from baseline in the patient assessment of the daily Average Hemophilic arthropathy Pain Intensity score on a 0- to 10-point numeric rating scale where 0 = no pain and 10 = pain as bad as you can imagine. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Judith Boice, PhD, Study Director — Tremeau Pharmaceuticals
Locations (45):
- United States (19):
  - Orthopedic Hospital DBA Orthopedic Hemophilia Treatment Center, Los Angeles, California
  - Center for Inherited Blood Disorders, Orange, California
  - UC Davis Children's Hospital, Sacramento, California
  - University of Colorado Hemophilia & Thrombosis Center, Aurora, Colorado
  - Georgetown University Hospital - Medstar, Washington D.C., District of Columbia
  - University of Florida - Shands, Gainesville, Florida
  - Clinical Trial Services, Corp, Miami, Florida
  - Anchor Medical Research, LLC, Miami, Florida
  - Rush University Medical Center, Chicago, Illinois
  - University of Iowa Hospitals & Clinics, Iowa City, Iowa
  - Louisiana Center for Bleeding and Clotting Disorders, New Orleans, Louisiana
  - Johns Hopkins University, Baltimore, Maryland
  - ECMC Hospital, Buffalo, New York
  - Icahn School of Medicine at Mount Sinai., New York, New York
  - East Carolina University, Greenville, North Carolina
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Oregon Health & Science University, Portland, Oregon
  - North Texas Comprehensive Hemophilia Center, Dallas, Texas
  - Gulf States Hemophilia and Thrombophilia Center, Houston, Texas
- Australia (3):
  - Calvary Mater Newcastle, Waratah, New South Wales
  - Fiona Stanley Hospital, Murdoch, Western Australia
  - The Alfred Hospital, Melbourne
- Canada (2):
  - Health Sciences Center, St. John's, Newfoundland and Labrador
  - Hamilton Health Sciences Centre, Hamilton, Ontario
- Italy (2):
  - Azienda Ospedaliera Universitaria Policlinico Sant'Orsola Malpighi, Bologna
  - Ospedale Pediatrico Bambino Gesù, Roma
- Poland (2):
  - Centrum Medyczne Pratia Poznan, Poznan
  - Uniwersytecki Szpital Kliniczny im. Jana Mikulicza-Radeckiego we Wroclawiu, Wroclaw
- Hospital Universitario Central de Asturias, Oviedo, Principality of Asturias, Spain
- Turkey (Türkiye) (7):
  - Acibadem Adana Hospital, Adana
  - Akdeniz University Medical Faculty, Antalya
  - Erciyes University Medical Faculty, Edirne
  - Gaziantep University Medical Faculty Sahinbey Educational Research Hospital, Gaziantep
  - Istanbul University Cerrahpasa - Cerrahpasa Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Ondokuz Mayis Univ. Med. Fac., Samsun
- Ukraine (9):
  - CI Dnipropetrovsk CMCH #4 of Dnipropetrovsk RC, Dnipro
  - CI of Healthcare Kharkiv City Clin Children's Hosp #16 Kharkiv NMU, Kharkiv
  - Communal Institution of Kyiv Regional Council Kyiv Regional Clinical Hospital, Kyiv
  - Kyiv CCH #9 City SPC of Diagnostics & Treatment of Patients with HP, Kyiv
  - Nat.Children Specialized Hosp.OKHMATDYT of the Ministry of Health of Ukraine, Kyiv
  - SI Institute of Blood Pathology and Transfusion Medicine of NAMSU, Lviv
  - M.V. Sklifosovskyi Poltava RCH Dept of Pulmonology HSEIU Ukrainian Medical Stomatological Academy, Poltava
  - CI of TRC Ternopil UH, Ternopil
  - CI Zaporizhzhya Regional Clinical Hospital of ZRC, Zaporizhzhya